CLINICAL TRIAL: NCT02553746
Title: Study of the Use of Ultrasound Scan for Lumbar Regional Anesthesia
Brief Title: Ultrasound for Neuraxial Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Georgios Kotsovolis, Doctor, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14073
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Lumbar Ultrasound
Keywords: Ultrasound; Spinal anesthesia; Epidural anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental)
  Interventions: Device: Detection of the puncture site by ultrasound scan of the lumbar spine.
- Landmarks (Active Comparator)
  Interventions: Procedure: Detection of the puncture site by identification of the landmarks.

INTERVENTIONS:
Device: Detection of the puncture site by ultrasound scan of the lumbar spine. — Neuraxial anesthesia will be performed to the patients after detection of the puncture site by ultrasound scan of the spine. The scanning will be performed as described by Arzola et al. The L3-L4 space will be identified by palpation and identification of the landmarks (Tuffier's line). The ultrasound probe will be placed perpendicular to the long axis of the spine. The spinous process will be identified (bright signal followed by dark triangular area). The probe will be moved to cephalad or caudal to identify the intervertebral space and when the best view of the ligamentum flavum is achieved two marks will be drawn on the skin: one at the center of the upper surface of the probe and one at the center of the right lateral vertical side of the probe. The intersection of the two landmarks will be the puncture site. The distance from the skin to the ligamentum flavum will be measured by the ultrasound caliper.
  Arms: Ultrasound
Procedure: Detection of the puncture site by identification of the landmarks. — Neuraxial anesthesia will be performed to the patients after detection of the puncture site by the identification of the landmarks. The L3-L4 space will be identified by palpation of the posterior iliac crests and the ideal intervertebral space will be selected after palpation of the spinous processes.
  Arms: Landmarks

SUMMARY:
The patients will be allocated to 2 groups: the ultrasound group and the palpation group. Ultrasound detection of the puncture site will be performed to the patients of the one group (group U). The puncture site will be determined by palpation of the landmarks at the patients of the other group (group L). The main purpose of the study is to determine if the ultrasound scan of the lumbar spine can facilitate spinal, epidural and combined spinal-epidural anesthesia, increase the success and decrease the complication rate of these techniques. The secondary purpose of the study is to evaluate if the lumbar ultrasound scan can be used to determine accurately the depth of the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* Surgery under spinal, epidural or combined spinal-epidural anesthesia.
* Surgery under general anesthesia and preoperative placement of epidural catheter for postoperative analgesia.
* ASA 1-3.

Exclusion Criteria:

* History of lumbar spinal surgery.
* Low back pain at the time of anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kotsovolis, Principal Investigator — 424 Army General Hospital of Thessaloniki
Locations (1):
- 424 Army General Hospital Department of Anesthesia, Thessaloniki, Greece

REFERENCES:
- [Background] Ali ME, Laurito CE. Ultrasound guidance for epidural catheter placement: a coming of age? J Clin Anesth. 2005 May;17(3):235-6. doi: 10.1016/j.jclinane.2005.02.002. No abstract available. PMID 15896595
- [Background] Arzola C, Davies S, Rofaeel A, Carvalho JC. Ultrasound using the transverse approach to the lumbar spine provides reliable landmarks for labor epidurals. Anesth Analg. 2007 May;104(5):1188-92, tables of contents. doi: 10.1213/01.ane.0000250912.66057.41. PMID 17456672
- [Background] Arzola C, Mikhael R, Margarido C, Carvalho JC. Spinal ultrasound versus palpation for epidural catheter insertion in labour: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jul;32(7):499-505. doi: 10.1097/EJA.0000000000000119. PMID 25036283
- [Background] Balki M. Locating the epidural space in obstetric patients-ultrasound a useful tool: continuing professional development. Can J Anaesth. 2010 Dec;57(12):1111-26. doi: 10.1007/s12630-010-9397-y. Epub 2010 Nov 11. English, French. PMID 21063818
- [Background] Balki M, Lee Y, Halpern S, Carvalho JC. Ultrasound imaging of the lumbar spine in the transverse plane: the correlation between estimated and actual depth to the epidural space in obese parturients. Anesth Analg. 2009 Jun;108(6):1876-81. doi: 10.1213/ane.0b013e3181a323f6. PMID 19448216
- [Background] Darrieutort-Laffite C, Bart G, Planche L, Glemarec J, Maugars Y, Le Goff B. Usefulness of a pre-procedure ultrasound scanning of the lumbar spine before epidural injection in patients with a presumed difficult puncture: A randomized controlled trial. Joint Bone Spine. 2015 Oct;82(5):356-61. doi: 10.1016/j.jbspin.2015.02.001. Epub 2015 Mar 9. PMID 25764916
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Ultrasound imaging facilitates localization of the epidural space during combined spinal and epidural anesthesia. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):64-7. doi: 10.1053/rapm.2001.19633. No abstract available. PMID 11172514
- [Background] Grau T, Leipold RW, Delorme S, Martin E, Motsch J. Ultrasound imaging of the thoracic epidural space. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):200-6. doi: 10.1053/rapm.2002.29239. PMID 11915069
- [Background] Grau T, Leipold RW, Fatehi S, Martin E, Motsch J. Real-time ultrasonic observation of combined spinal-epidural anaesthesia. Eur J Anaesthesiol. 2004 Jan;21(1):25-31. doi: 10.1017/s026502150400105x. PMID 14768920
- [Background] Grau T, Leipold RW, Horter J, Conradi R, Martin EO, Motsch J. Paramedian access to the epidural space: the optimum window for ultrasound imaging. J Clin Anesth. 2001 May;13(3):213-7. doi: 10.1016/s0952-8180(01)00245-8. PMID 11377160
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Efficacy of ultrasound imaging in obstetric epidural anesthesia. J Clin Anesth. 2002 May;14(3):169-75. doi: 10.1016/s0952-8180(01)00378-6. PMID 12031746
- [Background] Helayel PE, da Conceicao DB, Meurer G, Swarovsky C, de Oliveira Filho GR. Evaluating the depth of the epidural space with the use of ultrasound. Rev Bras Anestesiol. 2010 Jul-Aug;60(4):376-82. doi: 10.1016/S0034-7094(10)70046-5. English, Portuguese. PMID 20659609
- [Background] Hotta K. [Ultrasound-guided epidural block]. Masui. 2008 May;57(5):556-63. Japanese. PMID 18516882
- [Background] Karmakar MK, Li X, Ho AM, Kwok WH, Chui PT. Real-time ultrasound-guided paramedian epidural access: evaluation of a novel in-plane technique. Br J Anaesth. 2009 Jun;102(6):845-54. doi: 10.1093/bja/aep079. Epub 2009 Apr 27. PMID 19398454
- [Background] Liu SS, Ngeow JE, Yadeau JT. Ultrasound-guided regional anesthesia and analgesia: a qualitative systematic review. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):47-59. doi: 10.1097/AAP.0b013e3181933ec3. PMID 19258988
- [Background] Luo L, Ni J, Wu L, Luo D. Ultrasound-guided epidural anesthesia for a parturient with severe malformations of the skeletal system undergoing cesarean delivery: a case report. Local Reg Anesth. 2015 May 6;8:7-10. doi: 10.2147/LRA.S81696. eCollection 2015. PMID 25999759
- [Background] Nassar M, Abdelazim IA. Pre-puncture ultrasound guided epidural insertion before vaginal delivery. J Clin Monit Comput. 2015 Oct;29(5):573-7. doi: 10.1007/s10877-014-9634-y. Epub 2014 Oct 28. PMID 25348834
- [Background] Peng PW, Rofaeel A. Using ultrasound in a case of difficult epidural needle placement. Can J Anaesth. 2006 Mar;53(3):325-6. doi: 10.1007/BF03022227. No abstract available. PMID 16527803
- [Background] Perlas A, Chaparro LE, Chin KJ. Lumbar Neuraxial Ultrasound for Spinal and Epidural Anesthesia: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):251-60. doi: 10.1097/AAP.0000000000000184. PMID 25493689
- [Background] Piosik ZM, Helbo-Hansen S, Sprehn M. [Ultrasound-guided performance of labour epidural analgesia in a patient with thoracolumbar scoliosis]. Ugeskr Laeger. 2015 Jan 26;177(2A):102-3. Danish. PMID 25612990
- [Background] Rasoulian A, Lohser J, Najafi M, Rafii-Tari H, Tran D, Kamani AA, Lessoway VA, Abolmaesumi P, Rohling RN. Utility of prepuncture ultrasound for localization of the thoracic epidural space. Can J Anaesth. 2011 Sep;58(9):815-23. doi: 10.1007/s12630-011-9548-9. Epub 2011 Jun 23. PMID 21698508
- [Background] Schlotterbeck H, Schaeffer R, Dow WA, Touret Y, Bailey S, Diemunsch P. Ultrasonographic control of the puncture level for lumbar neuraxial block in obstetric anaesthesia. Br J Anaesth. 2008 Feb;100(2):230-4. doi: 10.1093/bja/aem371. PMID 18211995
- [Background] Shaikh F, Brzezinski J, Alexander S, Arzola C, Carvalho JC, Beyene J, Sung L. Ultrasound imaging for lumbar punctures and epidural catheterisations: systematic review and meta-analysis. BMJ. 2013 Mar 26;346:f1720. doi: 10.1136/bmj.f1720. PMID 23532866
- [Background] Singh S, Wirth KM, Phelps AL, Badve MH, Shah TH, Sah N, Vallejo MC. Epidural catheter placement in morbidly obese parturients with the use of an epidural depth equation prior to ultrasound visualization. ScientificWorldJournal. 2013 Jul 25;2013:695209. doi: 10.1155/2013/695209. eCollection 2013. PMID 23983645
- [Background] Taninishi H, Kawano K, Morita K. Ultrasound-assisted epidural anesthesia to amyotrophic woman. J Anesth. 2013 Oct;27(5):797-8. doi: 10.1007/s00540-013-1600-1. Epub 2013 Apr 2. No abstract available. PMID 23546640
- [Background] Vaghadia H, Germain G, Tang R. Epidural analgesia in parturients with ankylosing spondylitis: a role for ultrasound surveillance and ultrasound-guided placement. Can J Anaesth. 2013 Feb;60(2):206. doi: 10.1007/s12630-012-9822-5. Epub 2012 Nov 22. No abstract available. PMID 23180059
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Wang Q, Yin C, Wang TL. Ultrasound facilitates identification of combined spinal-epidural puncture in obese parturients. Chin Med J (Engl). 2012 Nov;125(21):3840-3. PMID 23106885
- [Background] Wight JM, Male D, Combeer A. Ultrasound-guided combined spinal-epidural anaesthesia for elective caesarean section in a patient with achondroplasia. Int J Obstet Anesth. 2013 Apr;22(2):168-9. doi: 10.1016/j.ijoa.2013.01.007. Epub 2013 Mar 7. No abstract available. PMID 23473550
- [Background] Yamashita J, Yamauchi M, Yamakage M. [Utility of ultrasound imaging for epidural blood patch in postdural puncture headache patients after caesarean section]. Masui. 2011 Jul;60(7):870-2. Japanese. PMID 21800673

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound: Detection of the puncture site by ultrasound scan of the lumbar spine.: Neuraxial anesthesia will be performed to the patients after detection of the puncture site by ultrasound scan of the spine. The L3-L4 space will be identified by palpation and identification of the Tuffier's line. The ultrasound probe will be placed perpendicular to the long axis of the spine. The spinous process will be identified. The probe will be moved to cephalad or caudal to identify the intervertebral space and when the best view of the ligamentum flavum is achieved two marks will be drawn on the skin: one at the center of the upper surface of the probe and one at the center of the right lateral vertical side of the probe. The intersection of the two landmarks will be the puncture site.
Period: Overall Study
Arm/Group | Ultrasound | Landmarks
Started | 80 | 66
Completed | 77 | 64
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound | Landmarks | Total
Number analyzed (Participants) | 80 | 66 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.42 (18.948) | 56.32 (19,961) | 54.24 (19.387)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 57 | 41 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 80 | 66 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 80 | 66 | 146
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.764 (3.784) | 28.427 (5.158) | 28.12 (4.5)
Type of anaesthesia [Count of Participants; unit: Participants]
  Spinal anaesthesia | 45 | 43 | 88
  Epidural anaesthesia | 9 | 7 | 16
  Combined spinal-epidural anaesthesia | 26 | 16 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Techniques
Description: For spinal and epidural anesthesia, success of the technique is defined as the installation of sensory block before surgery. For epidural catheter placement success of the technique is defined as the installation of sensory block after the end of surgery.
Time Frame: An expected average of 10 minutes after the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants | 74 | 63
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p = 0.748, Chi-squared, Corrected

2. Primary Outcome: Number of Participants With Success of the Technique at the First Attempt
Description: Number of patients with completion of the technique without any withdrawal or reposition of the needle.
Time Frame: An expected average of 10 minutes after the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants | 48 | 35
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p = 0.498, Chi-squared, Corrected

3. Primary Outcome: Number of Attempts Required.
Description: How many times did the operator withdraw the needle and repeated the puncture.
Time Frame: An expected average of 10 minutes after the technique..
Measure: Mean (Standard Deviation); unit: number of attempts
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
number of attempts | 1.65 (0.978) | 2.06 (1.413)
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p = 0.171, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Repositioning Frequency.
Description: How many times did the operator change the trajectory of the needle.
Time Frame: An expected average of 10 minutes after the technique.
Measure: Mean (Standard Deviation); unit: repositioning attempts
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
repositioning attempts | 0.74 (0.973) | 1.14 (1.357)
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p = 0.162, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Number of Participants With Change of the Intervertebral Space.
Description: Number of patients to whom the operator had to perform the puncture at a different intervertebral place than the initial one.
Time Frame: An expected average of 10 minutes after the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants | 14 | 20
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p = 0.104, Chi-squared, Corrected

6. Primary Outcome: Time Required.
Description: Time passed from the positioning of the patient on the table until the end of the neuraxial anesthesia
Time Frame: An expected average of 15 minutes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
seconds | 550.46 (214.016) | 451.94 (291.473)
Statistical Analysis 1: Comparison: Ultrasound vs Landmarks; Test type: Superiority; p < 0.005, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Depth of the Epidural Space Measured by Ultrasound.
Description: The distance between the skin and the ligamentum flavum measured by the built-in ultrasound caliper.
Time Frame: An expected average of 3 minutes after the beginning of the procedure.
Population: Data not collected
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Depth of the Epidural Space Measured by the Needle.
Description: The distance between the skin and the ligamentum flavum measured by the markers on the Tuohy needle.
Time Frame: An expected average of 5 minutes after the beginning of the procedure.
Reporting Status: Not Posted

9. Secondary Outcome: Number of Patients With Low Back Pain.
Description: Number of patients who reported low back pain after the technique.
Time Frame: 12hours and 24hours after the end of the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants | 11 | 11

10. Secondary Outcome: Low Back Pain Intensity.
Description: The patient is asked to evaluate the lumbar pain by the 11scale Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Time Frame: 12hours and 24hours after the end of the technique.
Population: Data not collected
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Patient Satisfaction.
Description: The patient is asked if he is satisfied with the technique (Definitely not, Not completely, Yes) and if he would choose the same technique in the future (Yes/No).
Time Frame: 12hours after the end of the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants
  Yes | 74 | 63
  Not exactly | 3 | 1
  No | 0 | 0

12. Secondary Outcome: Number of Participants With Any Complication.
Description: Number of patients who had any complication after the technique
Time Frame: 24hours after the end of the technique.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Landmarks
Number analyzed (Participants) | 77 | 64
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 24 hours after the completion of the technique
Description: The intervention of the study consists of ultrasound imaging which doesn't carry any risk for serious adverse events nor it can potentially affect all-cause mortality
Arm/Group | Ultrasound | Landmarks
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/66
Other Adverse Events (participants affected / at risk) | 80/80 | 66/66
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrasound (N=80) | Landmarks (N=66)
Skin irritation (Skin and subcutaneous tissue disorders) | 80 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT02553746/Prot_SAP_000.pdf